CLINICAL TRIAL: NCT05331313
Title: Analysis of Genomic Alterations in Sporadic Cases of Multiple Myeloma
Brief Title: The Aim is to Identify Recurrent Genomic Mutations and/or Predisposing Polymorphisms in Patients With Sporadic Cases of Multiple Myeloma
Acronym: MMSPORADGEN
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_0492
Record Dates: First submitted 2022-03-31; First posted 2022-04-15 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-03

CONDITIONS: Multiple Myeloma
Keywords: genetic predisposition; mutations; sporadic; multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Genetic Predisposition to Disease | interventions — Sequence Analysis, DNA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA analyses will be performed on purified abnormal plasmocytes, obtained from bone marrow aspirates performed during the standard follow-up of patients with multiple myeloma.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with a diagnosis of multiple myeloma: This study will involve a single patient group, namely patients with a diagnosis of multiple myeloma diagnosed by a bone marrow aspirate with cytological analysis of the bone marrow smear.Bone marrow samples obtained during the routine follow-up will undergo plasmocyte enrichment using immunopurification using CD138+ beads and nucleic acids will be extracted for sequencing.
  Interventions: Genetic: DNA sequencing

INTERVENTIONS:
Genetic: DNA sequencing — The aim of this study is to perform DNA sequencing on abnormal plasmocytes obtained from patients with multiple myeloma, in order to identify alterations which are associated with the existence of this disease. DNA analyses will be performed in a single experiment once all samples have been collected.

SUMMARY:
There is a growing body of data suggesting that the the risk of developing multiple myeloma, or myelomagenesis, is associated with genetic alterations occurring in the tumor cells. A limited number of candidate genes and polymorphisms have been reported in patients with this disease. In this study the investigators will compare the genetic information obtained on purified abnormal plasmocytes obtained from patients with multiple myeloma with available public databases in an effort to identify and if possible validate the role of certain mutations and/or polymorphisms in myelomagenesis. Plasmocytes will be obtained by immunomagnetic enrichment using CD138+ beads.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of multiple myeloma
* availability of abnormal plasmocytes

Exclusion Criteria:

- none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient samples will be accrued from Intergroupe Francophone du Myélome (IFM) centers in France, in the context of primary care clinics. The investigators aim to collect up to 1,000 samples.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
DNA mutations associated with the existence of multiple myeloma | baseline, pre-intervention/procedure/surgery
  DNA data acquired in myeloma patient samples will be compared to those of healthy subjects using publically available databases.
DNA mutations associated with the existence of multiple myeloma | during the intervention/procedure/surgery
  DNA data acquired in myeloma patient samples will be compared to those of healthy subjects using publically available databases.
DNA mutations associated with the existence of multiple myeloma | immediately after the intervention/procedure/surgery
  DNA data acquired in myeloma patient samples will be compared to those of healthy subjects using publically available databases.
DNA mutations associated with the existence of multiple myeloma | at 1 year
  DNA data acquired in myeloma patient samples will be compared to those of healthy subjects using publically available databases.
DNA mutations associated with the existence of multiple myeloma | up to 24 weeks
  DNA data acquired in myeloma patient samples will be compared to those of healthy subjects using publically available databases.
DNA mutations associated with the existence of multiple myeloma | through study completion, an average of 1 year
  DNA data acquired in myeloma patient samples will be compared to those of healthy subjects using publically available databases.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Pierre-Bénite, France